CLINICAL TRIAL: NCT04013893
Title: Evaluation of Enteral Nutrition in Critically Ill Children Receiving Inotropic Support in Pediatric Intensive Care Unit
Brief Title: Evaluation of Enteral Nutrition in Critically Ill Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ahmet Yontem, Principal Investigator, Cukurova University
Other Study IDs: CUTF-GOKAEK-86
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Critical Illness; Enteral Feeding Intolerance
Keywords: Enteral feeding; vasopressor; lactate
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to evaluate the effect of calorie and enteral feeding timing on survival in critically ill children receiving inotropic, vasopressor and inodilatory supplements.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of calorie and enteral feeding timing on survival in critically ill children receiving inotropic, vasopressor and inodilatory supplements. Early enteral nutrition will be initiated within the first 24 hours of hospitalization in critically ill children who have inotropic vasopressor and inodilator support without any problems and contraindications in gastrointestinal system functions. The energy requirement of the intubated patients will be measured by indirect calorie meter method. Schofield method will be used to calculate the daily energy needs of extubated patients. 30% of the targeted energy in the first 48 hours of hospitalization and 80% of the targeted energy in the first week will be achieved by enteral nutrition.Nutritional solutions with a concentrated formula of 1 / 1.5 will be given to patients with cardiac pulmonary or renal disease requiring fluid restriction.Patients will be followed up for vomiting, diarrhea, abdominal distention, feeding intolerance, gastric residues and gastrointestinal bleeding. If these findings develop, the patient's nutrition will be interrupted according to the clinician's assessment and enteral nutrition will be re-fed as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Children with normal gastrointestinal system function
* Children receiving inotropic, vasopressor or inodilatory support

Exclusion Criteria:

* Children with gastrointestinal system dysfunction
* Children with enteral nutrition contraindicated
* Children with metabolic disease with special nutrition

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill children who have inotropic, vasopressor or inodilatory supplements without any problems and contraindications in gastrointestinal system functions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
28-d mortality | 28 days
  To evaluate the effect of enteral feeding timing on survival

SECONDARY OUTCOMES:
Lactate | During inotropic treatment
  To observe safe lactate levels suitable for enteral nutrition. Lactate levels will be measure 4 times in a day.
Vasoactive inotrope score | During inotropic treatment
  To observe maximum vasoactive inotrope score suitable for enteral nutrition. Maximum VIS will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Dincer Yildizdaş, Professor, Study Chair — Cukurova University Medicine Faculty
Locations (1):
- Cukurova University, Division of Pediatric Intensive Care Unit, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided